CLINICAL TRIAL: NCT00472472
Title: Paclitaxel Coated Balloon Catheter for Inhibition of Restenosis in Femoropopliteal Arteries (PACCOCATH - FEM I)
Brief Title: Paclitaxel Coated Balloon Catheter for Prevention of Restenosis in Femoropopliteal Arteries
Acronym: PACCOCATH_F
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Charite Hospital, Berlin, Charite Hospital, Berlin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PACCOCATH - FEM I
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2007-05

CONDITIONS: Peripheral Arterial Disease
Keywords: restenosis; peripheral arterial disease; paccocath; drug-coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): PTA
  Interventions: Device: paclitaxel coated balloon catheter (device with drug)
- 2 (Active Comparator): PTA with Paccocath
  Interventions: Device: paclitaxel coated balloon catheter (device with drug)

INTERVENTIONS:
Device: paclitaxel coated balloon catheter (device with drug) — PTA vs Paccocath

SUMMARY:
The PACCOCATH FEM study is a randomized, double-blinded German multicenter trial on the efficacy and tolerance of a paclitaxel coated balloon catheter in prevention of restenosis after femoropopliteal angioplasty.

DETAILED DESCRIPTION:
Background: Treatment of patients with peripheral arterial disease (PAD) in the femoropopliteal arteries by percutaneous intervention is still limited by high rates of restenosis. The aim of the present study is to evaluate the efficacy and safety of a novel method of short time local drug delivery based on a paclitaxel-coated balloon in femoropopliteal arteries.

Methods and results: The double-blind and randomized study enrolled n=79 patients with occlusion or stenosis of femoropopliteal arteries. Inclusion criteria were clinical Rutherford stage 1-5, occlusion or hemodynamic relevant stenosis (≥ 70 % diameter) of femoropopliteal arteries and successful guiding wire recanalization. The primary endpoint was the late lumen loss after 6 months follow-up as seen in angiography. Secondary endpoints included the rate of restenosis (a binary variable), change of ankle brachial index (ABI), rutherford class and major adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford stage 1, 2, 3, 4 oder 5
* Occlusion or Stenosis of Superficial femoral and/or popliteal artery
* Successful guide wire passage of the lesion
* Patient suitable of vascular surgery in case of complication
* Written consent
* Patient is willing to take part in follow up examinations within the study

Exclusion Criteria:

* Acute ischemia
* Distal run off less than one vessel
* Pregnancy
* Hyperthyroidism
* Thrombocytes <100.000/mm3 or >700.000/mm3, Leucocytes <3.000/mm3
* Life expectancy less than two years
* Patients not willing to enter the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2004-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
angiographic late lumen loss | 6 months

SECONDARY OUTCOMES:
binary restenosis rate; major adverse events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ricke, MD, Principal Investigator — Klinik für Strahlenheilkunde, Charité Campus Virchow, Augustenburger Platz 1, 13353 Berlin, Germany; Ulrich Speck, PhD, Study Director — Radiologie, Campus Mitte, Charite, 10117 Berlin, Germany
Locations (2):
- Germany (2):
  - Klinik für Strahlenheilkunde, Charité Campus Virchow Klinikum, Berlin
  - Institut für Diagnostische Radiologie und Neuroradiologie, Universitätsklinikum Greifswald der Ernst-Moritz-Arndt-Universität, Greifswald

REFERENCES:
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Speck U, Scheller B, Abramjuk C, Grossmann S, Mahnkopf D, Simon O. Inhibition of restenosis in stented porcine coronary arteries: uptake of Paclitaxel from angiographic contrast media. Invest Radiol. 2004 Mar;39(3):182-6. doi: 10.1097/01.rli.0000116125.96544.64. PMID 15076010
- [Background] Scheller B, Speck U, Schmitt A, Bohm M, Nickenig G. Addition of paclitaxel to contrast media prevents restenosis after coronary stent implantation. J Am Coll Cardiol. 2003 Oct 15;42(8):1415-20. doi: 10.1016/s0735-1097(03)01056-8. PMID 14563585
- [Background] Scheller B, Speck U, Romeike B, Schmitt A, Sovak M, Bohm M, Stoll HP. Contrast media as carriers for local drug delivery. Successful inhibition of neointimal proliferation in the porcine coronary stent model. Eur Heart J. 2003 Aug;24(15):1462-7. doi: 10.1016/s0195-668x(03)00317-8. PMID 12909076
- [Background] Scheller B, Speck U, Bohm M. Prevention of restenosis: is angioplasty the answer? Heart. 2007 May;93(5):539-41. doi: 10.1136/hrt.2007.118059. PMID 17435062
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Speck U, Scheller B, Abramjuk C, Breitwieser C, Dobberstein J, Boehm M, Hamm B. Neointima inhibition: comparison of effectiveness of non-stent-based local drug delivery and a drug-eluting stent in porcine coronary arteries. Radiology. 2006 Aug;240(2):411-8. doi: 10.1148/radiol.2402051248. PMID 16864669
- [Derived] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447